CLINICAL TRIAL: NCT00242905
Title: Anatomical and Functional MRI Study of Episodic Memory in Epileptic Compared to Normal Children
Brief Title: Functional Magnetic Resonance Imaging (fMRI) Study of Memory in Children
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick VACHER, Department of Clinical Research of developpement
Other Study IDs: P040203
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2007-03

CONDITIONS: Childhood Absence Epilepsy [Pyknolepsy]
Keywords: Memory; Epilepsy; Children; Magnetic resonance imaging; Functional magnetic resonance imaging
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Study of memory using MRI — Study of memory using MRI

SUMMARY:
Memory is a cognitive function whose development is still poorly documented in children, but which is often disturbed in temporal epilepsy. There are no studies about the disorders of episodic memory. The investigations using functional MRI (fMRI) are scarce, they do not involve this field and none are dedicated to children. The objectives of this project are to study the neuronal networks involved in episodic memory in normal children, as well as the disorders of episodic memory in children with epilepsy and the mechanisms of cognitive and cerebral reorganization in epilepsy.

DETAILED DESCRIPTION:
Twenty children aged from 6 to 18 years with temporal and/or frontal epilepsy and 20 normal children in the same age range will undergo the following examinations in a unique day in the Unit Hospital F. JOLIOT(CEA in ORSAY, France):

1. complete neuropsychological evaluation including episodic memory,
2. structural MRI to quantify, using VBM, the potential abnormalities of the anatomical structures, to perform cognitive-morphological correlations, and to localize the neuronal networks activated on fMRI,
3. functional MRI using an original task of episodic memory, specifically dedicated to children and being under behavioural validation laboratory.

The analysis of fMRI data will be performed using SPM and taking into account the existence of epilepsy or not, of cerebral lesion or not, age, handedness, the side and location of epileptogenic focus, the age of seizure onset, and the type of antiepileptic treatment.

This study has been approved by the Ethic Committee in september 2004 (CCPPRB BICETRE, promotion of ASSISTANCE PUBLIQUE - HOPITAUX de PARIS).

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal tutors of the children having given written consent to participate to the study, after having being fully informed.
* Patients presenting with a temporal and/or frontal epilepsy and being able to perform the tasks of the protocol.
* Controls being recruited among brothers, sisters, and friends of the patients and being right-handlers, without any neurological history or learning disorders.

Exclusion Criteria:

* Any contra-indication to MRI or being claustrophobia or blind.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Inclusion Criteria:
  * Parents or legal tutors of the children having given written consent to participate to the study, after having being fully informed.
  * Patients presenting with a temporal and/or frontal epilepsy and being able to perform the tasks of the protocol.
  * Controls being recruited among brothers, sisters, and friends of the patients and being right-handlers, without any neurological history or learning disorders.
  Exclusion Criteria:
  * Any contra-indication to MRI or being claustrophobia or blind.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2005-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CHIRON, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Service Hospitalier Frédéric Joliot (SHFJ), Orsay
  - Necker Hospital, Paris

REFERENCES:
- [Background] Jambaque I, Dellatolas G, Dulac O, Ponsot G, Signoret JL. Verbal and visual memory impairment in children with epilepsy. Neuropsychologia. 1993 Dec;31(12):1321-37. doi: 10.1016/0028-3932(93)90101-5. PMID 8127430
- [Background] Hertz-Pannier L, Chiron C, Jambaque I, Renaux-Kieffer V, Van de Moortele PF, Delalande O, Fohlen M, Brunelle F, Le Bihan D. Late plasticity for language in a child's non-dominant hemisphere: a pre- and post-surgery fMRI study. Brain. 2002 Feb;125(Pt 2):361-72. doi: 10.1093/brain/awf020. PMID 11844736